CLINICAL TRIAL: NCT04582656
Title: Prospective Multicenter Trial Assessing the Efficacy of a Novel 3D Cartography-based Targeted Focal Microwave Therapy in Men With Localized Intermediate-risk Prostate Cancer
Brief Title: Efficacy Assessment of a Novel 3D Cartography-based Targeted Focal Microwave Therapy in Men With Localized Intermediate-risk Prostate Cancer
Acronym: VIOLETTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koelis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIOLETTE; 2019-A00803-54 (Other: ANSM)
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: Cancer; Prostate; Targeted treatment; Microwave
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicenter, single-arm, open-label, 12-month follow-up clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Targeted microwave ablation (Experimental): Targeted microwave transrectal or transperineal ablation of the prostatic index tumor using MRI-transrectal image registration and OBT fusion
  Interventions: Device: Targeted microwave ablation

INTERVENTIONS:
Device: Targeted microwave ablation — Targeted ablation of the index tumor with microwaves, by using either a transperineal or a transrectal approach

SUMMARY:
Multicenter, prospective, European, single-arm, open-label, 12-month follow-up clinical trial. The purpose of this study is to evaluate the efficacy of a 3D cartography-based targeted microwave ablation for the treatment of the index lesion in patients with intermediate risk prostate cancer.

DETAILED DESCRIPTION:
European and American guidelines recommend several therapeutic alternatives: radical surgical treatment, external beam radiotherapy or brachytherapy. However, whole-gland treatment induces significant morbidity and burden on quality of life. Targeted treatments of the index tumor are currently under investigation to decrease morbidity while proposing active treatment.

The purpose of this study is to assess the efficacy of a novel ablation treatment using microwaves, delivered transrectally or transperineally under real-time guidance with MRI-transrectal ultrasound image registration. The index tumor will be detected with prostate MRI and characterized with targeted biopsies using Organ Based Tracking (OBT) fusion with the TRINITY system (KOELIS, Meylan, France). The same system will be used to identify the index lesion and guide the targeted microwave ablation performed with the TATO3 device (Biomedical Srl, Florence, Italy).

All patients will undergo biopsy at 12 months of follow-up. A biopsy session will also be performed at 6 months, but only for patients with imaging results suspicious for cancer within the ablated area on the mpMRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 45 to 76 years old
* Life expectancy >10 years at the inclusion time
* Patient diagnosed with an intermediate-risk prostate cancer, defined by:

  * A T1c or T2a clinical stage
  * A unique cancer focus of Gleason (3+4) (Grade Group 2)
  * A PSA level <20 ng/mL
* Cancer focus identified on a multiparametric MRI of the prostate no more than 3 months before inclusion
* Confirmation of the suspicion of cancer identified on the MRI with transrectal or transperineal targeted and systematic biopsies performed with the KOELIS TRINITY system (no more than 3 months before inclusion)
* Patient suitable for IV sedation or general anesthesia and focal microwave ablation
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up
* Known coagulopathy or bleeding disorders are controlled
* Free, informed and written consent, dated and signed before the enrollment and before any exam required by the trial
* Patient affiliated to social security regimen or beneficiary of such regimen for local regions

Exclusion Criteria:

* Past medical history of prostate surgery
* Past medical history of radiotherapy or pelvic trauma
* Past medical history of acute prostatitis
* Presently taking hormonal manipulation or androgen supplements.
* Past medical history of cancer in the 5 previous years, excluding a non-metastatic basal cell carcinoma of the skin
* Severe BPH-related urinary tract symptoms, defined by an IPSS score >18
* Serious medical illness, including any of the following: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction, cerebrovascular event within 6 months prior to the screening visit
* Contraindications for MRI exam
* Extracapsular cancer extension or seminal vesicles or pelvic lymph node invasion suspected on prostate MRI
* Presence of two or more clinically significant cancer foci in the inclusion biopsy exam
* Presence of a clinically significant cancer with a Gleason score ≥8 (Grade Group ≥4)
* Tumor largest axis >12 mm on the prostate MRI
* Distance between the cancer focus and the apex <10 mm on the prostate MRI
* Distance between the cancer focus and the rectum <5 mm on the prostate MRI
* Patient already participating in an interventional clinical trial
* Patient protected by law

Ages: 45 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with no evidence of cancer on targeted biopsy | 12 months
  The proportion of patients with no evidence of cancer on targeted biopsy at 12 months, defined by a minimum of 2 targeted core biopsies taken from the index tumor site treated with microwave ablation for focal treatment of intermediate risk prostate cancer

SECONDARY OUTCOMES:
Proportion of radical salvage treatment | 12 months
  Proportion of patients undergoing radical salvage treatment of the index lesion
Time to radical salvage treatment | 12 months
  Time to radical salvage treatment of the index lesion
Proportion of patients with any cancer in the untreated area | 12 months
  Proportion of patients with any cancer in the untreated area, determined by a minimum 12 cores systematic biopsy
Proportion of patients undergoing treatment for cancer in the untreated area | 12 months
  Proportion of patients undergoing treatment for cancer in the untreated area and time to treatment
IPSS questionnaire | 7 days and 1, 6 and 12 months
  Changes in patients' reported outcome measures (PROMs) for urinary symptoms using IPSS score compared to baseline, score ranging from 0 to 35 (the higher the worse)
IIEF-5 questionnaire | 7 days and 1, 6 and 12 months
  Changes in patients' reported outcome measures (PROMs) for erectile function using IIEF-5 score compared to baseline, score ranging from 5 to 25 (the lower the worse)
MSHQ-EjD-SF questionnaire | 7 days and 1, 6 and 12 months
  Changes in patients' reported outcome measures (PROMs) for ejaculatory function and bother using MSHQ-EjD-SF score compared to baseline, score ranging from 1 to 15 (the lower the worse) for ejaculatory function and from 0 to 5 for bother/satisfaction (the higher the worse)
Urine flow | 7 days and 1, 6 and 12 months
  Change in urine flow, using a uroflowmeter compared to baseline
Adverse events | 12 months
  Number and severity of device and procedure related adverse events
Patient post-operative pain level | Treatment day-evaluated between 2 and 4 hours after the procedure
  Average patient post-operative pain level reported on a pain numeric rating scale, with a range from 0 (no pain) to 10 (worst pain ever)
Patient satisfaction | 1, 6 and 12 months
  Patient satisfaction with the microwave ablation procedure as determined by questionnaire (no score assigned)
Ease of the procedure | Day 1
  Ease of the procedure measured with a score chosen by the operator (1: easy, 2: moderate, 3: difficult)
Duration of the procedure and associated variables | Day 1
  Duration of the procedure and associated variables
PSA | 1, 3, 6, 9 and 12 months
  Change in PSA measurement compared to baseline
PSA Nadir | 12 months
  Time to PSA Nadir after treatment of the index lesion
Prostate volume | 7 days and 6 and 12 months
  Change in volume of the prostate on the mpMRI compared to baseline
Patient motivation | Baseline
  Characterization of patient motivation to undergo targeted microwave ablation for treatment of the index lesion, as assessed by patient questionnaire (no score assigned)

CONTACTS AND LOCATIONS:
Overall Officials: Roland VAN VELTHOVEN, MD, Study Chair — Uro Science & Consulting
Locations (7):
- Institut Jules Bordet, Brussels, Belgium
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hôpital de la Pitié-Salpêtrière (Assistance Publique - Hôpitaux de Paris), Paris
  - Hôpital Cochin (Assistance Publique - Hôpitaux de Paris), Paris
  - Urologie Nantes Clinique & Institut d'Urologie - Site Atlantis, Saint-Herblain
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No